CLINICAL TRIAL: NCT02769364
Title: Long-term Eribulin Treatment in Metastatic Breast Cancer: A Multicenter, Case-study Analysis
Brief Title: Extended Treatment in Metastatic Breast Cancer With Eribulin
Acronym: EXTER
Status: Completed | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: OBU-SW-H-05
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Advanced or Metastatic Breast Cancer; Eribulin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Participants treated with eribulin for at least 7 months

SUMMARY:
Decision-making for treatment of metastatic breast cancer after the second line of chemotherapy was limited by the lack of established predictive factors of benefit for further chemotherapy regimens. Eribulin has emerged as the only single agent demonstrating an overall survival improvement in the third-line setting or beyond. The purpose of this study was to define the clinical profile of metastatic breast cancer participants achieving long-term benefit from chemotherapy with eribulin in the third-line setting or beyond.

DETAILED DESCRIPTION:
This was a multicenter, retrospective, observational, case study analysis to assess long-term eribulin treatment in metastatic breast cancer. The study was conducted in 26 Spanish hospitals participating in a national pre-market access program to eribulin between 2011 and 2014. An exploratory comparison with a group of short-term responders included in a similar observational study was performed.

ELIGIBILITY:
Inclusion criteria:

* Participants with Advanced or Metastatic Breast Cancer on Eribulin for at least 7 months

Exclusion criteria:

* Lack of accessible clinical records

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Advanced or Metastatic Breast Cancer on Eribulin for at least 7 months
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 7 months
Progression free survival (PFS) | up to 7 months
Objective response rate | up to 7 months
Time to response | up to 7 months
Post progression survival | up to 7 months

SECONDARY OUTCOMES:
Number of participants with adverse events/serious adverse events/toxic deaths as a measure of safety | up to 7 months

CONTACTS AND LOCATIONS:
Locations (21):
- Spain (21):
  - Santiago de Compostela, A Coruña
  - Las Palmas de Gran Canarias, Gran Canaria
  - San Sebastián, Guipuzcoa
  - Barbastro, Huesca
  - Alcorcón, Madrid
  - Aravaca, Madrid
  - Pozuelo de Alarcón, Madrid
  - Pamplona, Navarre
  - Bilbao, Vizcaya
  - Badajoz
  - Cáceres
  - Jaén
  - Lleida
  - Madrid
  - Málaga
  - Murcia
  - Ourense
  - Salamanca
  - Seville
  - Valencia
  - Zaragoza